CLINICAL TRIAL: NCT04601844
Title: An Open-Label, Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Doses of Subcutaneously Administered Human Monoclonal Antibody Pozelimab in Combination With Single Doses of Subcutaneously Administered siRNA Cemdisiran in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Pozelimab in Combination With Cemdisiran in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3918-HV-1982; 2020-000300-11 (EudraCT Number)
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Cemdisiran at dose 1 SC single dose on day 1 followed by pozelimab at dose 1 SC single dose on day 29
  Interventions: Drug: Pozelimab; Drug: Cemdisiran
- Cohort 2 (Experimental): Cemdisiran at dose 2 SC single dose on day 1 followed by pozelimab at dose 1 SC single dose on day 29
  Interventions: Drug: Pozelimab; Drug: Cemdisiran
- Cohort 3 (Experimental): Cemdisiran at dose 2 SC single dose and pozelimab at dose 2 SC single dose, both administered on day 1
  Interventions: Drug: Pozelimab; Drug: Cemdisiran

INTERVENTIONS:
Drug: Pozelimab — Single dose administered subcutaneously
  Other Names: REGN3918
Drug: Cemdisiran — Single dose administered SC
  Other Names: ALN-CC5

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of ascending doses of subcutaneous (SC) pozelimab and SC cemdisiran when administered on the same day or sequentially 28 days apart.

The secondary objectives of the study are:

* To assess the concentration-time profiles of total pozelimab, total complement component 5 (C5), cemdisiran, and cemdisiran metabolite(s) following single ascending doses of SC pozelimab and SC cemdisiran when administered on the same day or sequentially 28 days apart
* To assess the pharmacodynamic (PD) profile of ascending doses of SC pozelimab and SC cemdisiran, as well as when administered on the same day or sequentially 28 days apart
* To assess the immunogenicity of pozelimab and cemdisiran

ELIGIBILITY:
Key Inclusion Criteria:

1. Has a body mass index less than 30 kg/m2 at the screening visit
2. Judged to be in good health as defined in the protocol
3. Is in good health based on laboratory safety testing obtained at the screening visit NOTE: Subject with a history of Gilbert's disease can be enrolled in the study
4. Willing to undergo vaccination against Neisseria meningitidis unless subjects have documentation of completed series of vaccinations within the past 2 years of the screening visit
5. Must have two negative COVID-19 tests taken 48 hours apart and within 7 days prior to study drug administration

Key Exclusion Criteria:

1. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or neurological disease, as assessed by the investigator that may confound the results of the study or poses an additional risk to the subject by study participation
2. Hospitalization (>24 h) for any reason within 30 days of the screening visit
3. Has a confirmed positive drug test result at the screening visit and/or prior to enrollment; or a history of recreational drug use (eg, marijuana) and/or drug or alcohol abuse within a year prior to the screening visit
4. Is positive for HIV, hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb), hepatitis C antibody and positive for qualitative (ie, detected) HCV RNA test at the screening visit
5. Within the previous 2 months of the screening visit has a history of bacterial, protozoal, parasitic or viral infection (including COVID-19) and/or persistent chronic or active recurring infection which requires treatment with antibiotics, antivirals, or antifungals
6. Known or suspected COVID-19 disease
7. Known allergy or intolerance to penicillin class antibiotics or macrolides

NOTE: Other protocol-defined Inclusion/ Exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) | Up to 20 weeks

SECONDARY OUTCOMES:
Concentrations of pozelimab in serum over time | Up to 20 weeks
Concentrations of cemdisiran in plasma over time | Up to 20 weeks
Concentrations of total C5 over time | Up to 20 weeks
Change from baseline in total complement hemolytic activity assay (CH50) over time | Up to 20 weeks
Incidence of treatment-emergent anti-drug antibodies (ADA) to pozelimab | Up to 20 weeks
Incidence of treatment-emergent anti-drug antibodies (ADA) to cemdisiran | Up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Regeneron Research Site, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/